CLINICAL TRIAL: NCT02547155
Title: Does Spinal Anesthesia for Prolapse Surgery With Concomitant Sling Procedures Lead to an Increase in Urinary Retention Compared to General Anesthesia?
Brief Title: Does Spinal Anesthesia for Prolapse Surgery With Lead to Urinary Retention?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Laura Martin, Urogynecology Fellow in the Department of Gynecology, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLA 15-019
Record Dates: First submitted 2015-07-15; First posted 2015-09-11 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Urinary Retention; Uterine Prolapse
MeSH Terms: conditions — Urinary Retention; Uterine Prolapse | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal anesthesia (Experimental): Subjects randomized to spinal anesthesia will receive Bupivacaine 0.75%, 8-12.5 mg dose depending on estimated duration of surgery and anesthesiologist decision. In addition to spinal anesthesia, these subjects will possibly have concurrent administration of fentanyl, midazolam, and propofol so that they are mildy sedated or sleeping.
  Interventions: Procedure: Spinal anesthesia
- General anesthesia (Active Comparator): Subjects randomized to general anesthesia will receive propofol induction, in combination with a muscle relaxant and inhalational gas per anesthesia standard of care at our institution
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Spinal anesthesia — 8-12.5 mg of bupivacaine will be administered for spinal anesthesia
  Arms: Spinal anesthesia
Procedure: General anesthesia — propofol induction, in combination with a muscle relaxant and inhalational gas
  Arms: General anesthesia

SUMMARY:
The purpose of the study is to compare the risk of being unable to urinate shortly after surgery, also called acute post-operative urinary retention (POUR) between spinal and general anesthesia in women who undergo outpatient pelvic organ prolapse with stress urinary incontinence surgery.

DETAILED DESCRIPTION:
A randomized trial to compare urinary retention rates between spinal and general anesthesia in women who undergo outpatient pelvic organ prolapse surgery with concomitant incontinence surgery.

Randomization

Randomization will be done in the pre-operative area, on the day of surgery. Computer generated randomization will be done in blocks of 4. Sealed numbered envelopes will be opened prior to surgery and the subject will then be assigned to spinal or general anesthesia. Patient randomization on day of surgery was discussed with anesthesia and it thought that randomizing on the same day would be safe.

Preoperatively

Subjects will be asked to complete a validated questionnaire, the Quality of Recovery 15 (QoR-15) prior to surgery, at their preoperative visit.

Anesthesia

Subjects randomized to general anesthesia will receive propofol induction, in combination with a muscle relaxant and inhalational gas per anesthesia standard of care at the investigators' institution.

Subjects randomized to spinal anesthesia will receive Bupivacaine 0.75%, 8-12 mg dose depending on estimated duration of surgery and anesthesiologist decision. In addition to spinal anesthesia, these subjects will possibly have concurrent administration of fentanyl, midazolam, and propofol so that they are mildy sedated or sleeping.

Voiding Trial

A voiding trial will be performed in the PACU once the subjects are able to stand and ambulate to the bathroom. Voiding trial will consist of removing the vaginal packing and back filling the bladder with 300cc of saline or less if subject has urgency or a smaller bladder capacity. A voiding trial is considered successful if the subject voids at least 2/3 of the total volume instilled and has a bladder scan showing less than 1/3 remaining. If a subject is unable to void after an hour, an additional hour will be permitted. However, after 2 hours from when the bladder was backfilled the subject is still unable to void, the Foley will be replaced and the subjects will be discharged home with a Foley leg bag and leg bag teaching.

An office nurse will call the subject and schedule an office nurse visit to remove the Foley between post-operative day number 5 to 7. If the subject goes home with a Foley this will be considered acute POUR.

Follow Up

Subjects will receive a phone call from either a nurse or fellow, between 48 to 72 hours post-operatively to make sure they are having no symptoms of urinary retention, are doing well and are not having any complications. A telephone survey will be administered during this follow up phone call using a validated questionnaire, the QoR-15. They will have received a copy of this survey to refer to at the time of their hospital discharge.

Subjects who were admitted to the hospital will have the same follow up, including a phone call 48 to 72 hours after their surgery, including the validated questionnaire, the QoR-15.

In addition, subjects will have a 6 week follow up visit in the clinic and will be asked to complete the QoR-15.

ELIGIBILITY:
Inclusion Criteria:

1. Women over the age of 40
2. Women scheduled for pelvic organ prolapse surgery as well as concomitant incontinence sling surgery
3. Post-void residual <150 cc prior to surgery
4. Surgery length of at least 1 hour
5. BMI <40
6. ASA class 1-2

Exclusion Criteria:

1. Contraindications to surgery
2. Contraindications to outpatient surgery, and requiring inpatient stay for medical comorbidities. The decision for a required inpatient stay will be decided prior to surgery based on the recommendations of the patient's primary care physician or specialist, such as cardiology or pulmonology.
3. BMI >40
4. ASA class 3 or 4 that would be a contraindiction to both spinal or general anesthesia
5. Evidence of voiding dysfunction or urinary retention on pre-operative urodynamics, including PVR >150, or dyssynergic sphincter dyssynergia
6. Neurological diseases that can interfere with spinal anesthesia
7. Anticoagulation therapy within a week of surgery
8. History of back surgery that would prevent successful spinal anesthesia
9. History of back deformity, such as scoliosis that would prevent successful spinal anesthesia

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative urinary retention | within the first week after surgery
  bladder emptying completeness after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Laura Martin, DO, Principal Investigator — Clevland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alas A, Martin L, Devakumar H, Frank L, Vaish S, Chandrasekaran N, Davila GW, Hurtado E. Anesthetics' role in postoperative urinary retention after pelvic organ prolapse surgery with concomitant midurethral slings: a randomized clinical trial. Int Urogynecol J. 2020 Jan;31(1):205-213. doi: 10.1007/s00192-019-03917-w. Epub 2019 Mar 23. PMID 30904934